CLINICAL TRIAL: NCT07339163
Title: Efficacy of Booster Injection With Gardasil-9 Vaccine on Intersurgical Interval (ISI) for Adults With Recurrent Respiratory Papillomatosis (RRP)
Brief Title: Efficacy of Booster Injection With Gardasil-9 Vaccine on Intersurgical Interval* for Adults With Recurrent Respiratory Papillomatosis*
Acronym: *ISI *RRP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Laura Matrka, Professor of Clinical Otolaryngology, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20251324
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Respiratory Papillomatosis (RRP)
Keywords: Recurrent Respiratory Papillomatosis (RRP); Human Papilloma Virus (HPV); Gardasil; Gardasil-9; Intersurgical Interval (ISI)
MeSH Terms: conditions — Recurrent respiratory papillomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Booster Administered (Experimental)
  Interventions: Biological: GARDASIL®9 (Human Papillomavirus 9-valent Vaccine, Recombinant)

INTERVENTIONS:
Biological: GARDASIL®9 (Human Papillomavirus 9-valent Vaccine, Recombinant) — Administration of Gardasil-9 vaccine as booster dose following 3-dose vaccine series in patients with RRP.

SUMMARY:
The investigators propose the study titled "Efficacy of booster injection with Gardasil-9 vaccine on intersurgical interval (ISI) for adults with recurrent respiratory papillomatosis (RRP)".

Recurrent respiratory papillomatosis (RRP) is a human papilloma virus (HPV) mediated disease of recurrent benign papillomas within the aerodigestive tract. While the foundation of treatment remains surgical debulking and occasionally adjuvant therapies such as cidofovir and bevacizumab, there remains a population of patients suffering from aggressive disease recurrence despite treatment.

Multiple studies have demonstrated treatment benefit in the form of an increase in intersurgical interval (ISI), following Gardasil vaccination. While adjuvant vaccination has favorably reduced recurrence of RRP and improved time course of disease recurrence for previously unvaccinated RRP patients, there remains a clinical population of adult patients suffering from persistent RRP that have previously undergone the Gardasil 3-vaccine series. Additionally, recent studies suggest a waning effect of Gardasil vaccination on ISI at longer time points.

Therefore, the investigators propose administering GARDASIL®9 (Human Papillomavirus 9-valent Vaccine, Recombinant) 0.5-mL suspension for injection as a one-time "booster" dose to adult patients >18 years of age, who have previously completed the 3-course vaccination series.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Has completed the 2- or 3-course Gardasil-9 vaccine series >2 years ago
3. Has a diagnosis of recurrent respiratory papillomatosis
4. Continue to have disease recurrence
5. Have at least 2 interventions (in order to calculate ISI)

Exclusion Criteria:

* Those who have not had at least two interventions prior to booster administration (inability to calculate ISI prior to 2- or 3-dose Gardasil-9 vaccine series and after completion of the vaccine series)
* Patients who have had no interventions for their disease since vaccination (unable to calculate post-Gardasil 2- or 3-dose vaccine series ISI)
* Have not completed the Gardasil-9 2- or 3-dose vaccine series greater than 2 years prior to proposed booster (not enough follow-up time to assess disease severity since vaccination)
* Patients with active any HPV-related cancer - their treatment course may impact the data collected during the study duration
* Any individual who has experienced anaphylaxis or hypersensitivity to a previous Gardasil vaccine (participation in this study would not be safe for the patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
Intersurgical Interval | 5 years
  The primary objective of this study is to compare the cohort-mean ISI-3 (post and the cohort-mean ISI-2 to assess whether ISI lengthens following booster administration. Our primary hypothesis is that administration of an additional booster shot of the Gardasil-9 vaccine in patients who have previously completed the 2- or 3-dose vaccine series will result in an increased ISI-3 as compared to ISI-2.
  The primary efficacy objective is to compare the cohort-mean of ISI-3 to the cohort-mean of ISI-2 to evaluate if administration of a booster dose of Gardasil-9 increases ISI. We will also calculate cohort-mean of ISI-1 to provide context and cohort ISI changes over time.
  Intersurgical Interval (ISI) - time, in days, between any two surgical interventions for treatment of a patient's disease ISI-1: ISI prior to the administration of the 2- or 3-dose Gardasil-9 course ISI-2: ISI before the booster Gardasil-9 dose, but after completion of the 2-or 3-dose course ISI-3: ISI post-booster
Safety and Adverse Events | 5 years
  The primary safety objective will characterize any adverse events and side effects that occur as a result of administration of the booster vaccine. Our primary safety hypothesis is that the administration of an additional booster vaccine of Gardasil-9 will not significantly increase the incidence of adverse events or side effects as compared to the side effect profile of the 2- or 3-dose vaccine series.

SECONDARY OUTCOMES:
Efficacy and Safety | 5 years
  Secondary objectives of this study are to further characterize the efficacy and safety of the Gardasil-9 booster in adults with recurrent respiratory papillomatosis (RRP) who have previously completed a 2- or 3-dose vaccine series. Specifically, we aim to evaluate the durability of ISI changes over time, assess subgroup differences (by age, sex, vaccination history, comorbidities, and baseline disease severity), and explore correlations between ISI improvement and key clinical outcomes such as recurrence rate and procedure frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Matrka, Doctor of Medicine, Principal Investigator — Ohio State University
Locations (1):
- Department of Otolaryngology - Head & Neck Surgery, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson EL, Freeman TE, Sun S, Koch B, Allen DZ, Sethia R, deSilva B, Matrka L. Recurrent respiratory papillomatosis disease course in immunosuppressed populations. J Laryngol Otol. 2024 May;138(5):576-580. doi: 10.1017/S0022215123001470. Epub 2023 Oct 25. PMID 37877153
- [Background] ."Census Profile: Columbus, OH Metro Area." Census Reporter, censusreporter.org/profiles/31000US18140-columbus-oh-metro-area/. Accessed 1 July 2024. "Health Equity." The Ohio State University Wexner Medical Center, wexnermedical.osu.edu/health-equity. Accessed 1 July 2024.
- [Background] Oshman LD, Davis AM. Human Papillomavirus Vaccination for Adults: Updated Recommendations of the Advisory Committee on Immunization Practices (ACIP). JAMA. 2020 Feb 4;323(5):468-469. doi: 10.1001/jama.2019.18411. No abstract available. PMID 31930397
- [Background] Buchinsky FJ, Ruszkay N, Valentino W, Derkay CS, McClay JE, Bastian RW, Myer CM, Lollar KW, Guris D. In RRP, serologic response to HPV is frequently absent and slow to develop. PLoS One. 2020 Mar 11;15(3):e0230106. doi: 10.1371/journal.pone.0230106. eCollection 2020. PMID 32160246
- [Background] Makiyama K, Hirai R, Matsuzaki H. Gardasil Vaccination for Recurrent Laryngeal Papillomatosis in Adult Men: First Report: Changes in HPV Antibody Titer. J Voice. 2017 Jan;31(1):104-106. doi: 10.1016/j.jvoice.2016.01.008. Epub 2016 Apr 8. PMID 27068425
- [Background] Tjon Pian Gi RE, San Giorgi MR, Pawlita M, Michel A, van Hemel BM, Schuuring EM, van den Heuvel ER, van der Laan BF, Dikkers FG. Immunological response to quadrivalent HPV vaccine in treatment of recurrent respiratory papillomatosis. Eur Arch Otorhinolaryngol. 2016 Oct;273(10):3231-6. doi: 10.1007/s00405-016-4085-3. Epub 2016 May 17. PMID 27188508
- [Background] Hocevar-Boltezar I, Maticic M, Sereg-Bahar M, Gale N, Poljak M, Kocjan B, Zargi M. Human papilloma virus vaccination in patients with an aggressive course of recurrent respiratory papillomatosis. Eur Arch Otorhinolaryngol. 2014 Dec;271(12):3255-62. doi: 10.1007/s00405-014-3143-y. Epub 2014 Jun 26. PMID 24964770
- [Background] Rosenberg T, Philipsen BB, Mehlum CS, Dyrvig AK, Wehberg S, Chirila M, Godballe C. Therapeutic Use of the Human Papillomavirus Vaccine on Recurrent Respiratory Papillomatosis: A Systematic Review and Meta-Analysis. J Infect Dis. 2019 Mar 15;219(7):1016-1025. doi: 10.1093/infdis/jiy616. PMID 30358875
- [Background] Ponduri A, Azmy MC, Axler E, Lin J, Schwartz R, Chirila M, Dikkers FG, Yang CJ, Mehta V, Gangar M. The Efficacy of Human Papillomavirus Vaccination as an Adjuvant Therapy in Recurrent Respiratory Papillomatosis. Laryngoscope. 2023 Sep;133(9):2046-2054. doi: 10.1002/lary.30560. Epub 2023 Jan 18. PMID 36651338
- [Background] Ivancic R, Freeman T, de Silva B, Forrest A, Kim B, Matrka L. Adjuvant Human Papillomavirus Vaccination in Recurrent Respiratory Papilloma Patients Older than 45. Laryngoscope. 2024 Jul;134(7):3226-3229. doi: 10.1002/lary.31368. Epub 2024 Feb 24. PMID 38401115
- [Background] Nyirjesy S, Osmundson P, Matrka L. Spontaneous Regression of Recurrent Respiratory Papillomatosis with HPV Vaccination: A Case Study. J Voice. 2022 Jul;36(4):587.e21-587.e25. doi: 10.1016/j.jvoice.2020.08.013. Epub 2020 Sep 3. PMID 32891477
- [Background] Ivancic R, Iqbal H, deSilva B, Pan Q, Matrka L. Current and future management of recurrent respiratory papillomatosis. Laryngoscope Investig Otolaryngol. 2018 Jan 14;3(1):22-34. doi: 10.1002/lio2.132. eCollection 2018 Feb. PMID 29492465
- [Background] Yiu Y, Fayson S, Smith H, Matrka L. Implementation of Routine HPV Vaccination in the Management of Recurrent Respiratory Papillomatosis. Ann Otol Rhinol Laryngol. 2019 Apr;128(4):309-315. doi: 10.1177/0003489418821695. Epub 2018 Dec 29. PMID 30595025
- [Background] Ballestas SA, Shelly S, Soriano RM, Klein A. Trends in recurrent respiratory papillomatosis treatment. Acta Otorrinolaringol Esp (Engl Ed). 2021 Mar-Apr;72(2):109-120. doi: 10.1016/j.otorri.2019.11.001. Epub 2020 Apr 17. English, Spanish. PMID 32312478